CLINICAL TRIAL: NCT03105999
Title: Observational Study On The Characterization Of 24-Hour Symptoms In Patients With COPD
Acronym: STORICO
Status: Completed | Type: Observational
Sponsor: Laboratori Guidotti S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: GUID/15/COPD/001
Record Dates: First submitted 2017-03-28; First posted 2017-04-10 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In COPD patients, a distinctive clustering of symptoms in the 3 parts of the day, early morning, day-time and night-time has been observed. These clusters are relevant to shape the health status and to explain the need of care. The objective of the STORICO study is to quantify the intra-day fluctuation of symptoms and to verify whether it: marks selected COPD phenotypes and is stable over time. STORICO is an observational prospective cohort multicenter study. 600 COPD patients >50 years will be enrolled. The multidimensional assessment will cover pattern of symptoms, complete spirometry and DLCO (Diffusing capacity of Lung for Carbon Monoxide ), comorbidity and health status. Based on clinical data, patients will be grouped in clinical phenotypes. Intra-day symptoms fluctuation will by rated by standardized questionnaires and the relationship between clinical/statistical clusters and symptoms fluctuations assessed. Finally, patients will be reassessed at 6 and 12 months, and the 12 month incidence of selected outcomes (frequency of exacerbations, use of health care resources) will be computed. Results are expected to clarify the classificatory and prognostic role of symptoms fluctuations in addition to classical measures of disease status and to compare health status and prognosis of clusters. Intra-day variations and stability of symptoms over time will likely improve our understanding of phenotypic variability of COPD.

DETAILED DESCRIPTION:
Primary objective - cross-sectional phase 1. To describe the frequency of early-morning, day- and night-time COPD symptoms according to phenotypes in a cohort of Italian patients with stable COPD (GOLD 2014 criteria). Symptoms will be evaluated by means of the Night-Time, Morning and Day-Time symptoms of COPD questionnaire. Primary objective - longitudinal phase 1. To describe the 12-month frequency and evolution of early-morning, day- and night-time COPD symptoms according to phenotypes measured at enrolment. Symptoms will be evaluated by means of the Night-Time, Morning and Day-Time symptoms of COPD questionnaire. Secondary objectives - cross sectional phase 1. To evaluate the association between early-morning, day- and night-time symptoms frequency at enrolment and the following outcomes: • dyspnea level • disease severity, as defined by the GOLD 2014 criteria (stages A to D) • quality of life • physical activity • quality of sleep • frequency and severity of exacerbations • level of depression and anxiety Secondary objectives - longitudinal phase 1. To describe the 12-month variation of the following outcomes according to phenotypes measured at enrolment: • dyspnea level • quality of life • physical activity • quality of sleep • frequency and severity of exacerbations • level of depression and anxiety 2. To describe the healthcare resources utilization in a cohort of Italian patients with COPD during 12-month observation, globally and by phenotypes. STUDY DESIGN: Italian observational cohort multicentre study in patients with stable COPD PLANNED NUMBER OF SUBJECTS: 600 patients STUDY PROCEDURE The study plan foresees: -Enrolment visit [Baseline visit (V1)] -A control visit at 6 months since Baseline at the investigational site (V2) -A final visit at 12 months since Baseline at the investigational site (V3) The clinical staff at the investigational sites will collect retrospectively all the necessary information about the medical history of the patient to confirm his-her eligibility. Patients confirmed with a diagnosis of stable COPD will be evaluated at enrolment visit and, if eligible, they will be asked to provide a written and signed privacy and informed consent form. The diagnosis of stable COPD should be compliant with 2014 GOLD criteria (stages A to D). At enrolment visit, patients will be asked to complete questionnaires for early-morning, day- and night-time symptoms, level of dyspnea, quality of life, physical activity, anxiety and depression levels, sleep quality, as well as to provide data on lifestyle, such as smoking. The investigator will be requested to complete study case report forms (CRFs) recording specified baseline information (demography data, medical history and comorbidities, COPD phenotype, ongoing treatments for COPD). Finally patients will perform a spirometry (baseline, lung volumes, bronchodilation test and CO diffusion) according to routine clinical practice. No additional mandated interventions on top of routinely performed physician visits, examinations or treatments will be required. Except the completion of the questionnaires, there are no other study-prescribed procedures. Any procedure ordered by the physician during this study will be one that is appropriate to the routine clinical care delivered to the COPD patients at the discretion of the physician. After 6 and 12 months, the same information as in the enrolment visits will be collected, excluding demographic data, to ascertain any changes in the outcomes of interest, including any exacerbations and medical healthcare resources utilization in the period between the visits. At follow up visits, patients will undergo the same procedures (spirometry) performed at the enrolment visit. For the entire period of observation, data regarding Adverse Event/Serious Adverse Event will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female outpatients aged ≥ 50
2. Diagnosis of stable COPD at least 12 months before the enrolment according to the GOLD 2014 criteria (stages A to D)
3. Current smokers or ex-smokers with a smoking history of ≥ 10 pack-years (e.g. 10 pack years = 1 pack /day x 10 years, or ½ pack/day x 20 years. An ex-smoker will be defined as a subject who has not smoked for ≥6 months at baseline)
4. Patients without any exacerbation at the baseline (enrolment visit) and in the last month prior to the enrolment visit
5. Patients must be able and willing to read and comprehend written instructions, and comprehend and complete the questionnaires required by the protocol
6. Patients who signed, after explanation, a written informed consent and privacy form, to confirm they understood the purpose of the study, and the procedure required in the study, and that they are willing to participate in the study.

Exclusion Criteria:

1. Patients participating in a clinical trial at enrolment
2. Patients who had changed active, dosage or frequency of administration of the maintenance therapy of COPD treatment regimen in the last 3 months prior to the enrolment visit (baseline)
3. Patients with a previous diagnosis of asthma, sleep apnea syndrome or other chronic respiratory disease different from COPD or other relevant medical conditions (on clinician's opinion) that will reduce the life expectancy of less than 3 years (Charlson index not including COPD >3)
4. Patients under long-term oxygen therapy

Study exit criteria:

1. Withdraw of informed consent to participate in the study
2. Diagnosis of asthma, sleep apnea syndrome or other chronic respiratory disease different from COPD
3. Death
4. Inclusion in a clinical trial

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with Pulmonary Disease, Chronic Obstructive
Sampling Method: Non-Probability Sample
Enrollment: 683 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2018-06-07 (Actual)

PRIMARY OUTCOMES:
Frequency of early-morning, day- and night-time COPD symptoms according to phenotypes in a cohort of Italian patients with stable COPD. Symptoms will be evaluated by means of the Night-Time, Morning and Day-Time symptoms of COPD questionnaire. | At baseline
  The frequency of early-morning, day and night-time symptoms at enrolment will be assessed based on the questions of the "Night-time, Morning and Day-time Symptoms of COPD questionnaire". It will be calculated within each class of phenotype as the ratio between the number of patients with at least 1 (early-morning, day and night-time) symptom in the week before enrolment and the total number of evaluable patients in the class. Three proportions will be calculated (for early-morning, day and night-time). The frequency of early-morning, day and night-time symptoms severity will be described too: for this reason, the proportion of mild, moderate, severe and very severe early-morning, day- and night-time symptoms in the week before enrollment will be provided.
  The frequency of specific COPD symptoms (breathlessness, coughing, bringing up phlegm or mucus, wheezing, chest tightness, chest congestion) will be also provided according to phenotypes.
12-month frequency and change from baseline of early-morning, day- and night-time COPD symptoms according to phenotypes measured at enrolment. Symptoms will be evaluated by means of the Night-Time, Morning and Day-Time symptoms of COPD questionnaire. | 6 and 12 months
  Phenotypes will be defined as per clinician judgment at enrollment. The proportion of patients changing phenotype during one-year observation provided.
  Within each class, the frequency of early-morning, day and night-time symptoms at each follow up visit will be calculated as the ratio between the number of patients with at least 1 symptom in the week preceding the follow up visit and the total number of evaluable patients in the class of phenotype with available "Night-time, Morning and Day-time Symptoms of COPD questionnaire" (COPD questionnaire) at follow up visit.
  For each patient the number of early-morning, day- and night-time symptom at each study visit together with the variation between visits will be calculated separately in the groups of patients according to baseline phenotype.
  The variation will be calculated as the difference between the number of symptoms at 12- (6-) month follow up and at baseline and between the number of symptoms at 12- and at 6-month follow up.

SECONDARY OUTCOMES:
Association between COPD symptoms frequency at enrolment and outcomes: • dyspnea level • disease severity (stages A to D GOLD 2014 criteria) • quality of life • physical activity • quality of sleep • exacerbations • depression and anxiety | At baseline
  The association at enrolment will be evaluated by calculating the frequency of symptoms in the groups of patients according to disease severity (A, B, C, D in GOLD 2014 guideline).
  Frequency of symptoms will be provided according to number of exacerbations in the year before baseline (0-1 vs ≥2) and to severity of exacerbations in the year before. Chi-squared tests (or Fisher exact tests if appropriate) will be provided too.
  The descriptive statistics of dyspnea level (mMRC score), quality of life (SGRQ symptoms, activity and impacts on daily life scores and total score), physical activity (IPAQ walking, moderate-intensity, vigorous-intensity activity and total scores), quality of sleep (CASIS total score), level of depression and anxiety (HADS anxiety, depression and total score) at enrollment in patients with vs without at least one symptom will be provided; the association between symptoms and outcomes will be evaluated by means of student T-test.
12-month variation of the following outcomes according to phenotypes measured at enrolment: • dyspnea level • quality of life • physical activity • quality of sleep • frequency and severity of exacerbations • level of depression and anxiety | 6 and 12 months
  At each follow up visit the following outcomes will be described and the variation (i.e. the difference) between each follow-up visit and since enrolment visit will be calculated by patient: dyspnea level (mMRC score), quality of life (SGRQ symptoms, activity and impacts on daily life scores and total score), physical activity (IPAQ walking, moderate-intensity, vigorous-intensity activity and total scores), quality of sleep (CASIS total score), level of depression and anxiety (HADS anxiety, depression and total score), number of exacerbations and of severe exacerbations. Such differences will be summarized by means of descriptive statistics globally and stratified by phenotype assessed at enrollment.
Healthcare resources utilization in a cohort of Italian patients with COPD during 12-month observation, globally and by phenotypes | 6 and 12 months
  The healthcare resources consumption will take into consideration the following events related both to management of COPD and to COPD exacerbations: inpatients and outpatients hospitalization, accesses to emergency department, GP and outpatient visits, laboratory tests, spirometry, pharmacological (LABA, LAMA, SABA, SAMA, etc.) and non-pharmacological therapies (rehabilitation) occurred/administered during study period.
  Medications for adverse events will be considered too. The annual direct healthcare resource consumption will be provided by means of descriptive statistics of the variables mentioned above.
  Analyses will be performed on the whole sample and stratified by phenotype.

CONTACTS AND LOCATIONS:
Locations (40):
- Italy (40):
  - Ospedale Ecclesiastico Miulli - Fisiopatologia Respiratoria, Acquaviva delle Fonti, Bari
  - A.O. Mellino Mellini - U.O. Fisiopatologia Respiratoria, Chiari, Brescia
  - Clinica Padre Pio - Medicina, Mondragone, Caserta
  - Ospedale Erba Renaldi - Medicina Interna, Menaggio, Como
  - Ospedale di Sestri Levante - Pneumologia, Sestri Levante, Genova
  - I.N.R.C.A. Centro per le Broncopneumopatie - Pneumologia Riabilitativa, Casatenovo, Lecco
  - Ospedale C. Cantù - Pneumologia, Abbiategrasso, Milano
  - Ospedale San Gerardo - Clinica Pneumologica, Monza, Monza E Brianza
  - Ospedale S. Maria della Pietà Camilliani - Pneumologia e Fisiologia Respiratoria, Casoria, Napoli
  - Ospedale Apicella - U.O.C. Pneumologia, Pollena Trocchia, Napoli
  - Ospedale Maggiore - U.O. Medicina, Modica, Ragusa
  - A.O.U. San Luigi Gonzaga - Malattie Apparato Respiratorio 1, Orbassano, Torino
  - Ospedale Civile - Pneumologia, Vittorio Veneto, Treviso
  - Ospedale di Dolo - U.O.C. Pneumologia, Dolo, Venezia
  - Ospedale INRCA - Clinica Medicina Interna e Geriatria, Ancona
  - Ospedale Cardinal G.Massaia - Pneumologia, Asti
  - A.O. San G.Moscati - U.O. Pneumologia, Avellino
  - Policlinico Consorziale - U.O. M.A.R., Bari
  - A.O. G.Rummo - U.O.C. Pneumologia, Benevento
  - Humanitas Gavazzeni - Pneumologia, Bergamo
  - A.O.U. Policlinico S.Orsola Malpighi - Pneumologia, Bologna
  - Policlinico Universitario Mater Domini - U.O.C. Malattie Apparato Respiratorio, Catanzaro
  - Ospedale Piero Palagi - Fisiopatologia Respiratoria e Riabilitazione Respiratoria, Florence
  - Ospedale D'Avanzo - MAR 4 Univ., Foggia
  - Ospedale Papardo - Malattie Apparato Respiratorio, Messina
  - A.O. San Carlo Borromeo - Pneumologia, Milan
  - Ospedale Niguarda - Pneumologia, Milan
  - A.O.U. Policlinico - Clinica Malattie Apparato Respiratorio, Modena
  - A.O.U. Seconda Università Napoli - UOSD Serv.Prevenz.Mal.Broncopolm., Napoli
  - Ospedale Zonchello - U.O.C. Pneumologia, Nuoro
  - Consiglio Nazionale delle Ricerche - Istituto di Biomedicina ed Immunologia Molecolare, Palermo
  - Fondazione Toscana G. Monasterio - U.O.C. Pneumologia, Pisa
  - Ospedale San Filippo Neri - U.O.C. Pneumologia, Roma
  - Ospedale Sandro Pertini - S.C. Pneumologia, Roma
  - Ospedale San Giovanni Addolorata - U.O.C. Malattie Apparato Respiratorio, Roma
  - Azienda Ospedaliera Sant'Andrea - U.O.C. Pneumologia, Roma
  - A.O.U. San Giovanni di Dio Ruggi d'Aragona - Pneumologia universitaria, Salerno
  - Ospedale Mazzini - Malattie Apparato Respiratorio, Teramo
  - Azienda Unità Sanitaria Locale Umbria n.2 - U.O. Pneumologia Terr., Terni
  - Ospedale Martini - Pneumologia, Torino

REFERENCES:
- [Background] Kessler R, Partridge MR, Miravitlles M, Cazzola M, Vogelmeier C, Leynaud D, Ostinelli J. Symptom variability in patients with severe COPD: a pan-European cross-sectional study. Eur Respir J. 2011 Feb;37(2):264-72. doi: 10.1183/09031936.00051110. Epub 2010 Nov 29. PMID 21115606
- [Background] Miravitlles M, Worth H, Soler Cataluna JJ, Price D, De Benedetto F, Roche N, Godtfredsen NS, van der Molen T, Lofdahl CG, Padulles L, Ribera A. Observational study to characterise 24-hour COPD symptoms and their relationship with patient-reported outcomes: results from the ASSESS study. Respir Res. 2014 Oct 21;15(1):122. doi: 10.1186/s12931-014-0122-1. PMID 25331383
- [Derived] Incalzi RA, Blasi F, Canonica GW, Foschino MP, Prediletto R, Simoni L, Ori A, Giovannetti C, Barsanti S, Scichilone N. The Prescribing Practice for COPD: Relationship to Circadian Rhythm, Disease Severity, and Clinical Phenotype in the STORICO Observational Study. Adv Ther. 2022 Dec;39(12):5582-5589. doi: 10.1007/s12325-022-02331-x. Epub 2022 Oct 11. PMID 36219388
- [Derived] Blasi F, Antonelli Incalzi R, Canonica GW, Schino P, Cuttitta G, Zullo A, Ori A, Scichilone N; STORICO study group. Clinical Evolution and Quality of Life in Clinically Based COPD Chronic Bronchitic and Emphysematous Phenotypes: Results from the 1-Year Follow-Up of the STORICO Italian Observational Study. Int J Chron Obstruct Pulmon Dis. 2021 Jul 21;16:2133-2148. doi: 10.2147/COPD.S310428. eCollection 2021. PMID 34345170
- [Derived] Antonelli Incalzi R, Canonica GW, Scichilone N, Rizzoli S, Simoni L, Blasi F; STORICO study group. The COPD multi-dimensional phenotype: A new classification from the STORICO Italian observational study. PLoS One. 2019 Sep 13;14(9):e0221889. doi: 10.1371/journal.pone.0221889. eCollection 2019. PMID 31518364
- [Derived] Scichilone N, Antonelli Incalzi R, Blasi F, Schino P, Cuttitta G, Zullo A, Ori A, Canonica GW; STORICO study group. Circadian rhythm of COPD symptoms in clinically based phenotypes. Results from the STORICO Italian observational study. BMC Pulm Med. 2019 Sep 9;19(1):171. doi: 10.1186/s12890-019-0935-2. PMID 31500607
- [Derived] Canonica GW, Blasi F, Scichilone N, Simoni L, Zullo A, Giovannetti C, Briguglio C, Barsanti S, Antonelli Incalzi R; STORICO study group. Characterization of circadian COPD symptoms by phenotype: Methodology of the STORICO observational study. Eur J Intern Med. 2017 Sep;43:62-68. doi: 10.1016/j.ejim.2017.05.021. Epub 2017 May 31. PMID 28576398
- See also: 1 Global Strategy for the Diagnosis, Management and Prevention of COPD, Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2014 — http://www.goldcopd.org